CLINICAL TRIAL: NCT00149370
Title: A Prospective Study of Patients Undergoing Breast Reduction Surgery: Health-Related Quality of Life and Clinical Outcomes
Brief Title: Quality of Life Among Breast Reduction Patients
Status: Completed | Type: Observational
Sponsor: Hamilton Health Sciences Corporation (Other)
Organization: McMaster University (Other)
Other Study IDs: 02-09-2005
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2005-09-08 (Estimated); Status verified 2005-08

CONDITIONS: Breast Hypertrophy
Keywords: breast hypertrophy; breast reduction surgery; health-related quality of life; Health Utilities Index; HUI; prospective; SF-36; quality-adjusted life years; QALY
MeSH Terms: conditions — Gigantomastia

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

INTERVENTIONS:
Procedure: Breast reduction surgery

SUMMARY:
Despite the growing evidence showing that breast hypertrophy is associated with reduced Health-Related Quality of Life (HRQL) and that reduction mammoplasty has a significant positive impact on HRQL, there are unresolved issues that need to be addressed. These include our ability to measure quantitatively the change that occurs after reduction and the ongoing restriction or denials of third party payments based on body mass index (BMI). The primary purpose of this study is to assess and measure the HRQL experienced by breast reduction patients using four reliable and validated HRQL measures.

Fifty-two consecutive patients with the diagnosis of breast hypertrophy were invited to participate in this prospective study. Participants completed the Health Utilities Index Mark 2 (HUI2) and Mark 3 (HUI3) and the Breast Reduction Assessment Value and Outcomes (BRAVO) instruments (the Short Form 36, the Multidimensional Body-Self Rating Questionnaire Appearance Assessment, and the Breast Related Symptom Questionnaire) at one week and one day pre-surgery and one, six, and 12 months post-surgery.

DETAILED DESCRIPTION:
This study addresses the following questions of clinical and policy relevance: 1) Is the pre-surgery HRQL of these patients compromised and, if so, in which areas? 2) Do patients' HRQL improve after surgery and, if so, when and in which areas and by how much? 3) Is there a relationship between BMI and pre-/post-surgery changes in HRQL (i.e., is the pre/post effect similar for both obese and non-obese patients)? and 4) Is there a relationship between tissue re-section weight and pre-/post-surgery changes in HRQL (i.e., is the pre/post HRQL effect similar for patients having small and large amounts of tissue resected)?

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of breast hypertrophy
* Government approval for payment of reduction mammoplasty

Exclusion Criteria:

* Unable or unwilling to complete the quality of life questionnaires

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52
Dates: Start 2001-01; Study Completion 2003-08

CONTACTS AND LOCATIONS:
Overall Officials: Achilleas Thoma, MD MSc FRCSC, Principal Investigator — McMaster Univeristy / St. Joseph's Healthcare
Locations (1):
- St. Joseph's Healthcare / McMaster University, Hamilton, Ontario, Canada

REFERENCES:
- [Result] Thoma A, Sprague S, Veltri K, Duku E, Furlong W. Methodology and measurement properties of health-related quality of life instruments: a prospective study of patients undergoing breast reduction surgery. Health Qual Life Outcomes. 2005 Jul 22;3:44. doi: 10.1186/1477-7525-3-44. PMID 16042775